CLINICAL TRIAL: NCT00490997
Title: A Prospective Randomized Double Blind Evaluation of Ketamine/Propofol vs Ketamine Alone for Pediatric Extremity Fracture Reduction
Brief Title: Ketamine/Propofol vs Ketamine Alone for Pediatric Fracture Reduction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-07-017; IRF 044-06
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2008-08

CONDITIONS: Fractures
Keywords: ketamine; propofol; sedation; pediatric; emergency department; fracture
MeSH Terms: conditions — Fractures, Bone; Emergencies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Ketamine only arm
  Interventions: Drug: Ketamine only
- 2 (Active Comparator): Ketamine-Propofol arm
  Interventions: Drug: Ketamine - Propofol

INTERVENTIONS:
Drug: Ketamine only — Ketamine 1.0 mg/kg IV and placebo intralipid as initial sedation agents (double blinded).
  Ketamine .25 mg/kg IV and placebo intralipid q2 minutes prn for additional sedation
  Arms: 1
Drug: Ketamine - Propofol — Ketamine .5 mg/kg and Propofol 1 mg/kg as initial sedation agents (double-blinded).
  Saline Placebo and Propofol .5 mg/kg q 2minutes for additional sedation
  Arms: 2

SUMMARY:
The objective of this study is to compare Ketamine-Propofol with Ketamine-only in a double-blind, randomised, controlled trial in a paediatric emergency department. We believe that the combination of these two agents will provide a new and more effective option for procedural sedation in paediatric emergency department patients. The hypothesis of the study is that paediatric emergency department patients requiring procedural sedation for an isolated orthopaedic injury with Ketamine-Propofol will have reduced total sedation time, time to recovery, complications and improved satisfaction scores compared to patients receiving Ketamine alone.

DETAILED DESCRIPTION:
Purpose: Procedural sedation has become an essential skill for emergency physicians, allowing for completion of painful procedures in a safe, comfortable and efficient manner. The ideal sedative agent would allow for an effective level of sedation, rapid onset and offset, absence of hemodynamic or respiratory compromise, and lack of post procedural side effects. A variety of agents have been studied for paediatric procedural sedation, however no currently used agent meets all of these criteria (1).

Background: Ketamine and Propofol are two agents that have been well studied and are commonly utilized as single agents for sedation. Ketamine is a dissociative agent that has amnestic and analgesic qualities. It has the unique property of allowing for deep sedation with minimal effects on the patient's respiratory drive. Ketamine use does not cause hypotension and in fact can have a positive effect on blood pressure. Ketamine has been extensively studied in paediatric sedation and has been found to be a safe and effective (2,3,4). Side effects associated with Ketamine use include post procedural nausea and vomiting, and unpleasant emergence phenomena such as agitation or hallucinations. Ketamine sedation can result in prolonged recovery times compared to other sedative agents and has a low rate of respiratory depression, apnea and laryngospasm (1).

Propofol is a sedative-hypnotic agent that has been popular for use in adult and paediatric procedural sedation for over a decade. The agent's rapid onset of effect and short duration of action allow for efficient sedation and recovery. Propofol has antiemetic properties and post-procedural side effects are rare. Caution must be used with Propofol, as it can be associated with significant respiratory depression and/or hypotension (1). The prolonged use of Propofol in children can produce acidosis, but this is not a problem for single use for an acute painful procedure.

A number of studies have demonstrated that the combination of Ketamine and Propofol for sedation is safe and effective, with most of the data in adults or in adult-child studies with small number of children (5,6). The combination of the two agents appears to reduce side effects of each medication used alone, and allows for a rapid recovery time. A prospective case series of Canadian emergency department patients given Ketamine-Propofol for procedural sedation has recently been published (5). In this study, 22% of the patients were children. However, to date there has been no targeted research published comparing Ketamine-Propofol head to head with any other presently utilized sedation regimen in a paediatric emergency department setting.

Objective & Hypothesis: The objective of this study is to compare Ketamine-Propofol with Ketamine-only in a double-blind, randomised, controlled trial in a paediatric emergency department. We believe that the combination of these two agents will provide a novel and more efficacious option for procedural sedation in paediatric emergency department patients. The hypothesis of the study is paediatric emergency department patients requiring procedural sedation for an isolated orthopaedic injury with Ketamine-Propofol will have reduced total sedation time, time to recovery, complications and improved satisfaction scores compared to patients receiving Ketamine alone.

Experimental Design: This study will be a prospective, double-blind, randomised, controlled clinical trial with an expected enrolment of approximately 140 patients from June-October 2007.

n = 2 * (Z1-α/2 + Z1-β)2 * σ2 / ∆2

n = 2 * (1.96 + 0.84)2 * 202 / 102

n = 2 * 7.84 * 400 / 100

n = 62.7 or 63 per group

Based on the calculation above, 63 children are needed in each group to have an 80% chance of detecting a clinically meaningful difference in total sedation time of 10 minutes between the groups, assuming an alpha of 0.05, and a standard deviation of 20 minutes. We have added an additional 7 patients (10%) to each group to account for potential drop-outs. Written, informed consent will be obtained from a parent/guardian for all children that meet the study inclusion criteria. Additionally, all children over the age of eight will also be asked for their assent.

Interventions: After giving informed consent, eligible patients will be assigned to either the Ketamine-Propofol group or Ketamine-placebo group through random allocation. Sealed envelopes containing a randomized assignment to either Ketamine-Propofol or Ketamine-only group will be prepared by an individual unconnected with the study using a web-based random number generator, balanced to ensure equal allocation to each group.

Patients in the Ketamine-only group will receive an intravenous dose of 1.0 mg/kg Ketamine and patients in the Ketamine-Propofol group will receive an intravenous dose of 0.5 mg/kg Ketamine and 1.0 mg/kg Propofol at time zero. Two minutes after the initial dose of sedative agent, and every 2 minutes thereafter, the attending physician will assess the patient's level of sedation using the Children's Hospital of Wisconsin Sedation Scale (Appendix A). If the attending physician determines the level of sedation is not adequate (Sedation score ≥ 3), additional study drugs (Ketamine group: 0.25 mg/kg Ketamine; Ketamine-Propofol group: 0.5 mg/kg Propofol) will be administered every 2 minutes until adequate sedation is achieved (deep conscious sedation = Children's Hospital of Wisconsin Sedation Scale Score < 3). Once a sedation score < 3 is achieved, the procedure will begin.

All sedation will be performed under continuous cardiorespiratory monitoring based on current hospital guidelines under the care and surveillance of a pediatric emergency department registered nurse and physician. Vital signs including heart rate, blood pressure, respiratory rate and oxygen saturation will be monitored continuously and recorded every 2 minutes, with the exception of blood pressure, which will be recorded every 4 minutes. The assisting registered nurse will also record information regarding time of last liquid and solid intake and body weight on the hospital's standard procedural sedation and analgesia record form.

A separate, standardized datasheet (Appendix B) will be used to collect the time when the study drug was first administered, the time when the procedure began, the time the procedure was completed and the time to recovery. Upon completion of the procedure, a recovery score based on a modified Aldrete Scale, will be recorded by a research associate blinded as to the intervention used every 2 minutes until full recovery, defined as a minimum cumulative score of 8. The attending physician will be asked to document any complications (including hypotension, apnea, hypoxia, laryngospasm and pain on injection) that occurred during the procedure and if any interventions were necessary. The nurse caring for the patient will also record any adverse events (nausea, vomiting, agitation) that occurred during recovery.

Outcome Measures: The primary outcome will be total sedation time, defined as the time that the first study drug was injected until the patient is fully recovered with a minimum recovery score ≥ 8. Secondary outcomes will include time to recovery; patient, nurse, and physician satisfaction; complications and adverse events. The patient, nurse and physician will be asked to individually assess their level of satisfaction with the sedation procedure using a 7-point Likert scale (Appendices C-E).

Analyses Strategy: The independent samples t-test will be used to compare differences in mean total sedation time and recovery time between the Ketamine and Ketamine-Propofol groups. The Mann-Whitney test will be used to compare differences in satisfaction levels (measured on an ordinal scale) between groups. Differences in proportions of complications during the procedure and adverse events during recovery will be assessed by the Chi-Square test between groups. A p value <0.05 will be considered statistically significant.

Expectation: The expectation of the study is paediatric emergency department patients requiring procedural sedation for an isolated orthopaedic injury with Ketamine-Propofol will have reduced total sedation time, time to recovery, complications and improved satisfaction scores compared to patients receiving Ketamine alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pediatric emergency patients with isolated extremity injury requiring reduction

Exclusion Criteria:

* Active respiratory illness
* Seizure disorder
* Craniofacial abnormalities
* Allergy to soy, ketamine, or propofol
* Hypertension
* Significant renal, cardiovascular or neurologic disease

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Total Sedation Time | defined as the time that the first study drug was injected until the patient is fully recovered with a minimum recovery score ≥ 8

SECONDARY OUTCOMES:
Time to Recovery | defined as the time interval from the last study drug given to recovery score ≥ 8
patient, nurse, and physician satisfaction | during and immediately after sedation
complications and adverse events | during and immediately after sedation

CONTACTS AND LOCATIONS:
Overall Officials: Amit P Shah, MD FCFP(EM), Principal Investigator — Western University, Canada; Greg Mosdossy, MD, FRCPC, Principal Investigator — Western University, Canada; Michael J Rieder, MD PhD FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- Children's Hospital of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Krauss B, Green SM. Procedural sedation and analgesia in children. Lancet. 2006 Mar 4;367(9512):766-80. doi: 10.1016/S0140-6736(06)68230-5. PMID 16517277
- [Background] Willman EV, Andolfatto G. A prospective evaluation of "ketofol" (ketamine/propofol combination) for procedural sedation and analgesia in the emergency department. Ann Emerg Med. 2007 Jan;49(1):23-30. doi: 10.1016/j.annemergmed.2006.08.002. Epub 2006 Oct 23. PMID 17059854
- [Background] Roback MG, Wathen JE, MacKenzie T, Bajaj L. A randomized, controlled trial of i.v. versus i.m. ketamine for sedation of pediatric patients receiving emergency department orthopedic procedures. Ann Emerg Med. 2006 Nov;48(5):605-12. doi: 10.1016/j.annemergmed.2006.06.001. Epub 2006 Aug 14. PMID 17052563
- [Background] Godambe SA, Elliot V, Matheny D, Pershad J. Comparison of propofol/fentanyl versus ketamine/midazolam for brief orthopedic procedural sedation in a pediatric emergency department. Pediatrics. 2003 Jul;112(1 Pt 1):116-23. doi: 10.1542/peds.112.1.116. PMID 12837876
- [Background] Cravero JP, Blike GT, Beach M, Gallagher SM, Hertzog JH, Havidich JE, Gelman B; Pediatric Sedation Research Consortium. Incidence and nature of adverse events during pediatric sedation/anesthesia for procedures outside the operating room: report from the Pediatric Sedation Research Consortium. Pediatrics. 2006 Sep;118(3):1087-96. doi: 10.1542/peds.2006-0313. PMID 16951002